CLINICAL TRIAL: NCT00180869
Title: A Randomized Study of Unmodified Versus Leuko-Reduced Allogeneic Red Blood Cells Transfusion During Surgery in Cancer Patients
Brief Title: Unmodified Versus Leuko-Reduced Allogeneic Red Blood Cells Transfusion in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANSFUGE
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Cancer; Surgery
Keywords: cancer; peroperative transfusion; allogeneic red blood cell concentrate; leuko-reduced red blood cell concentrate
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Procedure: transfusion of allogeneic red blood cell concentrate
Procedure: transfusion of leuko-reduced red blood cell concentrate

SUMMARY:
There is evidence to suggest that red blood cell concentrate (RBC) transfusion may have immunomodulatory effects. The aim of this randomized single-center trial is to compare immune responses in patients undergoing cancer surgery and given either an unmodified RBC (UN-RBC) or a leuko-reduced RBC (LR-RBC) transfusion perioperatively.

DETAILED DESCRIPTION:
This single-center study is conducted to compare the effect of peroperative transfusion of allogeneic unmodified RBC (UN-RBC) versus leuko-reduced RBC (RED-RBC) on recipient immunity. Patients undergoing cancer surgery are randomly assigned peroperatively to receive UN-RBC or RED-RBC. Groups are stratified for age, sex, tumor characteristics, prior transfusion and prior cancer treatment. Blood sampless are collected before anesthesia (d0) and at days 3, 7, 14 , 28 after transfusion/surgery and analyzed for complete cell blood count, lymphocyte subsets, cytokine production (IL4, IL10, IFNgamma, IL12), T-cells repertoire (TCR) analysis and detection of circulating donor cells. Main study endpoint is the influence of the treatment arm on IL4/IFNgamma ratio. The effect of transfusion type on any given biological parameters is also tested (peripheral blood mononuclear cell phenotyping (PBMC), cytokine production by stimulated PBMC, T cell repertoire analysis and microchimerism assessment).

ELIGIBILITY:
Inclusion Criteria:

* Surgery for cancer with a transfusion during surgery risk greater than 30%
* Surgery in curative intent
* Written informed consent

Exclusion Criteria:

* contraindications to the use of allogeneic unmodified red blood cell concentrate
* any anti-RBC and/or anti-HLA and/or anti-granulocyte alloimmunization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1997-09

PRIMARY OUTCOMES:
Polarization of lymphocyte responses towards a Th2 response following transfusion during surgery as assessed by the IL-4/IFN-γ ratio

SECONDARY OUTCOMES:
Peripheral blood mononuclear cell phenotyping
Cytokine production
Microchimerism at day 3 after transfusion during surgery
Alteration of T cell repertoire
Incidence of nosocomial infection
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lapierre, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France